CLINICAL TRIAL: NCT02498470
Title: Prospective Registry to Assess the Cath Lab Percutaneous Coronary Intervention Long-term Outcomes: a Single Center
Acronym: PCI-registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xiao-dong Zhuang (Other)
Responsible Party: Sponsor-Investigator, Xiao-dong Zhuang, diretor of the department of cardiology, the first affiliated hospital of sun yat-sen university, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: PCI-registry
Record Dates: First submitted 2015-07-12; First posted 2015-07-15 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: percutaneous coronary intervention — All the patients receiving coronal artery angiography or percutaneous coronary intervention therapy by standard protocol

SUMMARY:
The registry study is to obtain the state of the percutaneous coronary intervention state treatment for coronary heart disease in the center of the first hospital of sun yat-sen unversity in a real world.

DETAILED DESCRIPTION:
The registry study is to obtain the long-term outcomes of the percutaneous coronary intervention state treatment for coronary heart disease patients in the center of the first hospital of sun yat-sen unversity in a real world. The data are collected using an uploading system through internet.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving coronal artery angiography or percutaneous coronary intervention therapy

Exclusion Criteria:

* none

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients receiving coronal artery angiography or percutaneous coronary intervention therapy in the first affiliated hospital of sun yat-sen university
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2008-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Composite Major Adverse Cardiac Events (MACE) | 5 years
  All death All death, myocardial infarction, revascularization

SECONDARY OUTCOMES:
Target Lesion Failure | 5 year
  composite target lesion failure (TLF) defined as a composite of cardiac death, non-fatal myocardial infarction (MI) not clearly attributable to a nontarget vessel, or target lesion revascularization (TLR) (percutaneous or by coronary artery bypass grafting)

CONTACTS AND LOCATIONS:
Overall Officials: zhimin du, MD, Principal Investigator — first affiliated hospital of sun yat-sen university
Locations (1):
- Xiaodong Zhaung, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No